CLINICAL TRIAL: NCT06819410
Title: A Retrospective Clinical Study on the Efficacy and Safety of Amphotericin B Compared With Azoles in the Treatment of Invasive Fungal Disease
Brief Title: Efficacy and Safety of Amphotericin B and Azoles in the Treatment of Invasive Fungal Disease
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Deputy Chief Physician, Sichuan Provincial People's Hospital
Other Study IDs: Lunshen(Research)No.818,2024
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Invasive Fungal Disease
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment with polyene antifungal drugs: The dosage and course of Amphotericin B or Amphotericin B cholesteryl sulphate complex were determined by clinicians, and this study was registered according to clinical practice
- Treatment with azole antifungal drugs: The dosage and course of triazoles or imidazole antifungal drugs were determined by clinicians, and this study was registered according to clinical practice

SUMMARY:
Efficacy and safety of amphotericin B and azoles in the treatment of invasive fungal disease

DETAILED DESCRIPTION:
The medical records, demographic characteristics and clinical data of patients with invasive fungal disease treated with amphotericin B or azoles were collected through the electronic medical record system of Sichuan Provincial People's Hospital from 2021 to 2024. To evaluate the efficacy and safety of these two types of drugs.

ELIGIBILITY:
Inclusion Criteria:

* There is no age limit, gender is not limited
* Patients with invasive fungal disease who are treated with polyene antifungals or azole antifungals should be treated for ≥ 7 days.

Exclusion Criteria:

* Patients with incomplete data or other factors affecting the clinical outcome judgement
* Patients who are judged by the investigator to be unsuitable to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with invasive fungal disease who are treated with polyene antifungals or azole antifungals should be treated for ≥ 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | The end of treatment, up to 1 year
  Clinical success incudes cure or symptom improvement，which means patients are alive, IFD-related symptoms and signs, radiographic abnormalities improve or disappear completely, and microbiological evidence suggests fungal clearance. The proportion of patients with cured or improved symptoms in the total population was analyzed.

SECONDARY OUTCOMES:
Safety of amphotericin B and azoles | During the treatment (1-14 days); the end of treatment (Day 14);Day 28 after the start of treatment
  Safety evaluation was mainly based on the incidence of adverse events / adverse reactions in the two groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: lingai PP Pan, PhD, Study Chair — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No